CLINICAL TRIAL: NCT05426564
Title: Exploratory Assessment of the Quantra® System With the QPlus® and QStat® Cartridges in Adult ECMO Patients
Brief Title: Exploratory Assessment of the Quantra® System in Adult ECMO Patients
Status: Completed | Type: Observational
Sponsor: HemoSonics LLC (Industry)
Collaborators: University of California, Irvine (Other)
Responsible Party: Sponsor
Other Study IDs: HEMCS-041
Record Dates: First submitted 2022-06-07; First posted 2022-06-22 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Blood Loss; Thrombosis; Extracorporeal Circulation; Complications
Keywords: Quantra; ECMO; QPlus; Viscoelastic testing; Coagulation
MeSH Terms: conditions — Hemorrhage; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ECMO Patients: Patients undergoing an ECMO procedure
  Interventions: Diagnostic Test: Quantra System

INTERVENTIONS:
Diagnostic Test: Quantra System — Diagnostic device to monitor coagulation properties of a whole blood sample at the point-of-care.

SUMMARY:
This is a prospective, observational exploratory study of the performance of the Quantra System in adult patients that are undergoing an arterio-venous (AV), veno-venous (VV) ECMO or extra-corporeal life support (ECLS) procedure.

DETAILED DESCRIPTION:
Patients 18 years or older that are undergoing an arterio-venous (AV), veno-venous (VV) ECMO or extra-corporeal life support (ECLS) procedure will be enrolled in this prospective, observational exploratory study. From each enrolled subject, blood samples will be collected at multiple time points for analysis on the Quantra QPlus or QStat Cartridge in parallel with other assessments performed as standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Subject is > 18 years.
* Subject is scheduled to undergo either VA or VV ECMO procedure or has been placed on VA or VV ECMO within 24 hours.
* Subject or subject's legally authorized representative (LAR) is willing to provide informed consent, either prospectively or by deferred consent.

Exclusion Criteria:

* Subject is younger than 18 years of age.
* Subject is pregnant.
* Subject is incarcerated at the time of the study.
* Subject, or subject's legally authorized representative is unable or unwilling to provide informed consent.
* Subject is affected by a condition that, in the opinion of the treatment team, may pose additional risks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing arterio-venous (AV), veno-venous (VV) ECMO or extra-corporeal life support (ECLS) procedure. Both COVID-19 and non-COVID-19 related ECMO patients will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Comparison of Quantra Clot Time results to standard coagulation test results. | At the start of ECMO (considered the Baseline timepoint)
  Coagulation function assessed by Quantra and standard-of-care coagulation tests
Comparison of Quantra Clot Stiffness results to standard coagulation test results. | At the start of ECMO (considered the Baseline timepoint)
  Coagulation function assessed by Quantra and standard-of-care coagulation tests
Comparison of Quantra Clot Time results to standard coagulation test results. | 6 hours after the previous measurment
  Coagulation function assessed by Quantra and standard-of-care coagulation tests
Comparison of Quantra Clot Stiffness results to standard coagulation test results. | 6 hours after the previous measurment
  Coagulation function assessed by Quantra and standard-of-care coagulation tests

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Irvine, Irvine, California, United States